CLINICAL TRIAL: NCT04272346
Title: The Effects of Prosocial Writing on Psychological Well-being: An Online Randomized Controlled Trial Among Young Adult Cancer Survivors
Brief Title: Harnessing Generativity Among Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Marcie D. Haydon, MA, CPhil, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB# 19-001945
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cancer; Young Adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer helping condition (Experimental): Participants in the peer helping condition will be asked to write about their cancer experience with an emphasis on using the experience to benefit a newly-diagnosed AYA cancer patient.
  Interventions: Behavioral: Writing for others
- Processing + peer helping condition (Experimental): Participants in the processing + peer helping condition will be asked to first write about their deepest thoughts and feelings about their cancer experience (3 writings), then share advice to a newly-diagnosed AYA cancer patient (final writing).
  Interventions: Behavioral: Processing + writing for others
- Facts-only writing condition (Placebo Comparator): Participants in the facts-only writing condition will be asked to write about their cancer experience. Unlike the previous conditions, they will not be instructed to write for the benefit of a newly-diagnosed AYA cancer patient.
  Interventions: Behavioral: Facts-only writing

INTERVENTIONS:
Behavioral: Writing for others — Participants will receive general instructions for completing the writing sessions and will be asked to write for at least 20 minutes per session. Topics covered in each session will vary and are related to common cancer-related themes (e.g., receiving a diagnosis, undergoing treatment, etc.). Participants will be instructed not to worry about grammar, spelling, or sentence structure and reminded that their responses will remain anonymous. Writing sessions (four in total) will be spaced 1 week apart, and participants will be instructed to write about their experience for the benefit of a newly-diagnosed cancer patient.
  Arms: Peer helping condition
Behavioral: Processing + writing for others — Participants will receive general instructions for completing the writing sessions and will be asked to write for at least 20 minutes per session. Topics covered in each session will vary and are related to common cancer-related themes (e.g., receiving a diagnosis, undergoing treatment, etc.). Participants will be instructed not to worry about grammar, spelling, or sentence structure and reminded that their responses will remain anonymous. Writing sessions (four in total) will be spaced 1 week apart. For the first three writing sessions, participants will write their deepest thoughts and feelings regarding cancer diagnosis and treatment. In the final writing session, participants will be instructed to write about their experience for the benefit of a newly-diagnosed cancer patient.
  Arms: Processing + peer helping condition
Behavioral: Facts-only writing — Participants will receive general instructions for completing the writing sessions and will be asked to write for at least 20 minutes per session. Topics covered in each session will vary and are related to common cancer-related themes (e.g., receiving a diagnosis, undergoing treatment, etc.). Participants will be instructed not to worry about grammar, spelling, or sentence structure and reminded that their responses will remain anonymous. Writing sessions (four in total) will be spaced 1 week apart. Unlike the previous conditions, participants will not be instructed to write about their experience for the benefit of a newly-diagnosed cancer patient.
  Arms: Facts-only writing condition

SUMMARY:
Short, online interventions designed to enhance well-being may be particularly amenable for use with adolescent and young adult (AYA) cancer survivors (age 15-39 at diagnosis), an understudied group in the cancer community. The benefits of psychological well-being on both physical and mental health outcomes are well-known and, in recent years, researchers and policymakers have begun to view the period of adolescence and young adulthood as a window of opportunity to instantiate lasting habits and behaviors. Growing evidence suggests that prosocial behavior-a behavior that can be reliably manipulated through a short online intervention-may have beneficial effects on well-being and physical health. This has yet to be tested in AYA cancer survivors.

Drawing from the literature on positive psychology and prosocial interventions, the proposed study will test the feasibility and efficacy of an 8-week online peer helping intervention designed to increase well-being among AYA cancer survivors. AYA cancer survivors (n = 176) will be recruited and randomized to one of three conditions: a peer helping condition, a cancer-specific writing plus peer helping condition, or a cancer-specific writing condition (control condition). The second group was added in response to a previous study, which found that writing about one's experience prior to helping other survivors may be more beneficial. Participants will complete a weekly writing activity once per week for 4 weeks, with instructions administered via a weekly email. Participants will also complete online assessments before, during, and after the 4-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cancer (any type) between the ages of 15 and 39 years
* have completed primary treatment and are in remission (partial or complete)
* between the ages of 18 and 39 years
* fluent in English
* have access to the internet and email.

Exclusion Criteria:

-none

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Change in psychological well-being | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Well-being within the past month will be measured at baseline, post-intervention, and the 1-month follow-up via the 14-item Mental Health Continuum-Short Form (MHC-SF). The MHC-SF is comprised of three empirically derived subscales: the 3-item Emotional Well-Being Subscale, the 6-item Psychological Well-Being Subscale, and the 5-item Social Well-Being Subscale. Higher scores on each subscale, and the total score overall (range: 0-56), indicate greater well-being.

SECONDARY OUTCOMES:
Change in depressive symptoms | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Depressive symptoms over the past week will be measured at baseline, post-intervention, and the 1-month follow-up via the 20-item Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a measure of symptom severity, with higher scores (range: 0-60) indicating greater depressive symptoms.
Change in anxiety | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Symptoms of anxiety over the past 2 weeks will be measured at baseline, post-intervention, and the 1-month follow-up via the 7-item Generalized Anxiety Disorder- 7 (GAD-7). Higher scores on the GAD-7 (range: 0-21) indicate greater severity of symptoms.
Change in perceived impact of cancer | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Perceived impact of cancer will be measured at baseline, post-intervention, and the 1-month follow-up via the Impact of Cancer Scale, Version 2. The following subscales will be administered: positive self-evaluation (4 items; range: 4-20), worry (7 items; range: 7-35), body change concerns (3 items; range: 3-15), physical appearance concerns (3 items; range: 3-15), and altruism/empathy (4 items; range: 4-20. Higher scores on each subscale indicate greater perceived severity of impact.
Change in health-related quality of life | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Health-related quality of life over the past week will be measured at baseline, post-intervention, and the 1-month follow-up via 12-item Short Form Health Survey (SF-12). Higher scores on the SF-12 (range: 0-100) indicate greater quality of life.
Change in pain intensity and interference | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Pain intensity over the past week will be measured at baseline, post-intervention, and the 1-month follow-up using the 1-item PROMIS pain intensity questionnaire (range: 1-5). Pain interference over the past week will be measured at baseline, post-intervention, and the 1-month follow-up using the 4-item PROMIS pain interference questionnaire (range: 4-20). Higher scores indicate greater pain intensity and interference.
Change in cognitive functioning | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Cognitive functioning over the past week will be measured at baseline, post-intervention, and the 1-month follow-up using the 4-item PROMIS Cognitive Functioning Questionnaire (range: 4-20). Higher scores indicate greater cognitive functioning.
Change in sleep quality and disturbance | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Sleep quality and disturbance over the past week will be measured at baseline, post-intervention, and the 1-month follow-up using the 4-item PROMIS Sleep Disturbance Questionnaire (range: 4-20). Higher scores indicate greater sleep disturbance.
Change in fatigue | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Fatigue over the past week will be measured at baseline, post-intervention, and the 1-month follow-up using the 4-item PROMIS Fatigue Questionnaire (range: 4-20). Higher scores indicate greater fatigue.
Change in social support | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Social support will be measured at baseline, post-intervention, and the 1-month follow-up using the 21-item 2-way Social Support Scale. This scale measures 4 dimensions of social support: instrumental support received, instrumental support given, emotional support received, and emotional support given. A higher total score (range: 0-105) indicates more feelings of perceived support.
Change in generativity | At the baseline survey (the day the intervention begins), at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Feelings of generativity will be measured at baseline, post-intervention, and the 1-month follow-up using the 13-item Generativity Scale. This measure consists of two subscales: generative desire and generative achievement, with higher scores (range: 13-78) indicating greater desire/achievement.
Change in positive and negative affect | At the baseline survey (the day the intervention begins), at each writing session, at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Reports of positive and negative affect will be assessed at baseline, post-intervention, the 1-month follow-up, and at each writing session using the 10-item positive affect subscale and 10-item negative affect subscales of the Positive and Negative Affect Schedule (PANAS-X). Two additional adjectives were also included, happy and calm. Greater scores indicate higher feelings of positive (range: 10-50) and negative affect (range: 10-50).
Change in fulfillment of psychological needs | At the baseline survey (the day the intervention begins), at each writing session, at the post-intervention survey (1 week after the final writing assignment), and at the 1-month follow-up
  Fulfillment of psychological needs will be measured at baseline, post-intervention, the 1-month follow-up, and at each writing session using the 9-item Balanced Measure of Psychological Needs. This item has three subscales: autonomy, connectedness, and relatedness, with higher scores (range: 9-45) indicating greater needs satisfaction.

OTHER OUTCOMES:
Prosocial Tendencies (Moderator) | At the baseline survey (on the day of the first writing activity)
  Frequency of engaging in prosocial acts will be measured at baseline using the 20-item Self-Report Altruism Scale. Higher scores (range: 20-100) indicate more engagement in prosocial acts (e.g., helping a classmate with an assignment).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haydon MD, Stanton AL, Hoyt MA, Bower JE. A randomized controlled trial testing the benefits of prosocial writing in young adult survivors of adolescent and young adult cancer. Health Psychol. 2025 Sep;44(9):886-897. doi: 10.1037/hea0001512. Epub 2025 May 5. PMID 40323828